CLINICAL TRIAL: NCT06038331
Title: Evaluation of the Treatment of Symptomatic Scaphotrapeziotrapezoidal (STT) Osteoarthritis With a Treated, Devitalized and Sterile Amniotic Membrane of Umbilical Cord Placed in Joint Interposition
Brief Title: Use of a Treated, Devitalized and Sterile Umbilical Cord Amniotic Membrane in the Treatment of STT Osteoarthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SclerFIX-STT-TBF; 2023-A00790-45 (Other: IDRCB)
Record Dates: First submitted 2023-09-04; First posted 2023-09-14 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis Hand
Keywords: ScaphoTrapezioTrapezoid OsteoArthritis (STT OA)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SclerFIX-IP (Experimental): Treated, devitalised and sterile graft of umbilical cord amniotic membrane
  Interventions: Biological: SclerFIX-IP

INTERVENTIONS:
Biological: SclerFIX-IP — Decellularized, viro-inactivated, freeze-dried and sterile allogeneic graft of amniotic membrane of umbilical cord used as an interposition implant in the STT joint

SUMMARY:
The aim of this open, prospective, multicenter trial is to evaluate the use of a sterile, devitalized, processed umbilical cord amniotic membrane implant placed in joint interposition in the treatment of STT osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; age between 18 and 75 years.
* Patient with symptomatic STT OA.
* Patient treated medically for functional signs for more than 3 months, without improvement, justifying a surgical intervention.
* Patient with a QuickDash score > 33 points (converted to 50%).
* Patient with wrist pain in front of the STT joint at rest = or > 4/10 on VAS.
* Patient who received the study information and provided consent.
* Member or beneficiary of a national health insurance plan.

Exclusion Criteria:

* Pregnant or breastfeeding woman; woman without effective contraception.
* Patient with functional rhizarthrosis that has not been stabilized or treated medically or surgically.
* Patient with signs of neuropathy with functional disorders such as hyperesthesia.
* Patient with uncontrolled epilepsy or neuropathy that contraindicates locoregional anesthesia.
* Person confined by a judicial or administrative decision.
* Adult subjected to legal protection measures or unable to provide his/her consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Decrease of the symptomatology related to the STT OA | 12 months
  Quality of life related to STT OA evaluated using Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire (0 = no disability, 100 = most severe disability); a decrease of 25% of the score is expected between subject's inclusion and the 12-month postoperative visit

SECONDARY OUTCOMES:
Absence of inflammatory reactions and good local tolerance of the implant | Through study completion (12 months)
  No inflammatory reactions (oedema, erythema, necrosis, ulceration and/or delayed wound healing), no adverse effects or serious adverse effects.
Decrease of pain related to STT OA | 1 month, 3 months, 6 months, 12 months
  Pain evaluated from 0 (no pain) to 10 (worst imaginable pain) on a visual analog scale (VAS)
Improvement of functional activities involving the thumb | 1 month, 3 months, 6 months, 12 months
  Functional activities involving the thumb evaluated from 0 (best) to 56 (worst) using the Buffet score developed by the Besançon University Hospital
Increase of thumb strength | 3 months, 6 months, 12 months
  Thumb strength measured in kg by two-point pinch strength test using a pinch gauge
Increase of grip strength | 3 months, 6 months, 12 months
  Grip strength measured in kg by grip strength test using a dynamometer
No apparent joint space anomaly | 12 months
  Joint space evaluated on radiography using Crosby's classification

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Besançon, Besançon
  - Institut Chirurgical de la Main et du Membre Supérieur (ICMMS), Lyon
  - Centre de la Main - Clinique Jules Verne, Nantes
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No